CLINICAL TRIAL: NCT04222972
Title: A Phase III, Randomized, Open-Label Study of Pralsetinib Versus Standard of Care for First-Line Treatment of RET Fusion-Positive, Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Pralsetinib Versus Standard of Care for First-Line Treatment of Advanced Non-Small Cell Lung Cancer (NSCLC)
Acronym: AcceleRET-Lung
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO42864; 2019-002463-10 (EudraCT Number); BLU-667-2303 (Registry Identifier: CT.Gov); 2023-505035-12-00 (Other: EU CT number)
Expanded Access: NCT04204928 (Approved for marketing)
Record Dates: First submitted 2020-01-03; First posted 2020-01-10 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: RET-fusion Non Small Cell Lung Cancer; Lung Neoplasm; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Disease; Carcinoma, Bronchogenic; Bronchial Diseases; Head and Neck Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Germ Cell and Embryonal; Neoplasms, Nerve Tissue
Keywords: Advanced Non-Small Cell Lung Cancer; RET Lung; RET Mutation; RET Alteration; RET Positive; RET Inhibitor; RET Altered; RET Rearrangement; RET NSCLC; RET-Rearranged NSCLC; RET Fusion; RET Fusion Lung Cancer; M918T; TRIM33-RET; Lung Cancer Mutation; BLU 667; Pralsetinib; RET Tyrosine Kinase; RET Gene Mutation; RET Kinase; Advanced Lung Cancer; Metastatic Lung Cancer; KIF5B-RET; CCDC6-RET
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Bronchogenic; Bronchial Diseases; Head and Neck Neoplasms; Adenocarcinoma; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Germ Cell and Embryonal; Neoplasms, Nerve Tissue | interventions — pralsetinib; Carboplatin; Cisplatin; Pemetrexed; pembrolizumab; Gemcitabine; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pralsetinib (Experimental): Participants randomized to the Experimental Arm will receive Pralsetinib
  Interventions: Drug: Pralsetinib
- Platinum-based chemotherapy with or without pembrolizumab (Active Comparator): Participants randomized to the Active Comparator Arm will receive 1 of 6 platinum-based chemotherapy treatment regimens (with or without pembrolizumab) at the study center as chosen by the treating Investigator (based on histology)
  Nonsquamous histology
  * Carboplatin or cisplatin / pemetrexed (with vitamin supplementation); with optional pemetrexed (with vitamin supplementation) maintenance.
  * Pembrolizumab / carboplatin or cisplatin / pemetrexed (with vitamin supplementation); followed by pembrolizumab and optional pemetrexed (with vitamin supplementation) maintenance.
  Squamous histology
  * Carboplatin or cisplatin / gemcitabine
  * Carboplatin with paclitaxel/nab-paclitaxel and pembrolizumab
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Pemetrexed; Drug: Pembrolizumab; Drug: Gemcitabine; Drug: Paclitaxel; Drug: Nab-Paclitaxel

INTERVENTIONS:
Drug: Pralsetinib — Administered orally
  Other Names: BLU-667
  Arms: Pralsetinib
Drug: Carboplatin — Administered IV
  Arms: Platinum-based chemotherapy with or without pembrolizumab
Drug: Cisplatin — Administered IV
  Arms: Platinum-based chemotherapy with or without pembrolizumab
Drug: Pemetrexed — Administered IV
  Arms: Platinum-based chemotherapy with or without pembrolizumab
Drug: Pembrolizumab — Administered IV
  Arms: Platinum-based chemotherapy with or without pembrolizumab
Drug: Gemcitabine — Administered IV
  Arms: Platinum-based chemotherapy with or without pembrolizumab
Drug: Paclitaxel — Administered IV
  Arms: Platinum-based chemotherapy with or without pembrolizumab
Drug: Nab-Paclitaxel — Administered IV
  Arms: Platinum-based chemotherapy with or without pembrolizumab

SUMMARY:
This is an international, randomized, open-label, Phase 3 study designed to evaluate whether the potent and selective RET inhibitor, pralsetinib, improves outcomes when compared to a platinum chemotherapy-based regimen chosen by the Investigator from a list of standard of care treatments, as measured primarily by progression free survival (PFS), for participants with RET fusion-positive metastatic NSCLC who have not previously received systemic anticancer therapy for metastatic disease.

ELIGIBILITY:
Inclusion criteria:

* Participant has pathologically confirmed, definitively diagnosed, locally advanced (not able to be treated with surgery or radiotherapy) or metastatic NSCLC and has not been treated with systemic anticancer therapy for metastatic disease.
* Participant must have a documented RET-fusion
* Participant has measurable disease based on RECIST 1.1 as determined by the local site Investigator/radiology assessment.
* Participant has an ECOG Performance Status of 0 or 1.
* Participant should not have received any prior anticancer therapy for metastatic disease.

  * Participants can have received previous anticancer therapy (except a selective RET inhibitor) in the neoadjuvant or adjuvant setting but must have experienced an interval of at least ≥ 6 months from completion of therapy to recurrence.
  * Participants that received previous immune checkpoint inhibitors in the adjuvant or consolidation following chemoradiation are not allowed to receive pembrolizumab if randomized in Arm B
* Participant is an appropriate candidate for and agrees to receive 1 of the Investigator choice platinum-based chemotherapy regimens if randomized to Arm B.
* For women of childbearing potential: participants who agree to remain abstinent (refrain from heterosexual intercourse) or use contraception.
* For men: participants who agree to remain abstinent (refrain from heterosexual intercourse) or use a condom and agree to refrain from donating sperm.

Exclusion criteria:

* Participant's tumor has any additional known primary driver alterations other than RET, such as targetable mutations of EGFR, ALK, ROS1, MET, and BRAF. Investigators should discuss enrollment with Sponsor designee regarding co-mutations.
* Participant previously received treatment with a selective RET inhibitor.
* Participant received radiotherapy or radiosurgery to any site within 14 days before randomization or more than 30 Gy of radiotherapy to the lung in the 6 months before randomization.
* Participant with a history of pneumonitis within the last 12 months.
* Participant has CNS metastases or a primary CNS tumor that is associated with progressive neurological symptoms or requires increasing doses of corticosteroids to control the CNS disease. If a participant requires corticosteroids for management of CNS disease, the dose must have been stable for the 2 weeks before Cycle 1 Day 1.
* Participant has had a history of another primary malignancy that has been diagnosed or required therapy within the past 3 years prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Estimated at up to 32 months
  Defined as the time from randomisation date to the first documented progressive disease (PD), as assessed by investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Estimated at up to 32 months
  Defined as the proportion of participants who achieve a confirmed complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart, as assessed by investigator according to RECIST 1.1.
Overall Survival (OS) | Estimated at approximately 32 months
  Defined as the time from randomisation date to death due to any cause.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline, at every 21 day cycle visit until progressive disease or death (estimated 32 months)
  The intensity of Adverse Events (AEs) will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE v5.0).
Changes in Eastern Cooperative Oncology Group Performance Status (ECOG PS) | Baseline, at every 21 day cycle visit until progressive disease or death (estimated 32 months)
  Further characterising safety and tolerability.
Duration of Response (DOR) | Estimated at up to 32 months
  Defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as assessed by investigator according to RECIST v1.1.
Clinical Benefit Rate (CBR) | Estimated at up to 32 months
  Defined as the proportion of participants who experience a best response of Stable Disease (SD) with a minimum duration of 6 months, a CR, or a PR, as assessed by investigator according to RECIST v1.1.
Disease Control Rate (DCR) | Estimated at up to 32 months
  Defined as the proportion of participants who experience a best response of CR, or PR, or SD, as assessed by investigator according to RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (68):
- Hospital Britanico, Buenos Aires, Argentina
- Royal North Shore Hospital, St Leonards, New South Wales, Australia
- UZ Antwerpen, Edegem, Belgium
- Brazil (2):
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital A. C. Camargo, São Paulo, São Paulo
- Clinica CIMCA, San José, Costa Rica
- France (10):
  - Institut Bergonie CLCC Bordeaux, Bordeaux
  - Hôpital Ambroise Paré - Boulogne-Billancourt, Boulogne-Billancourt
  - CHRU Lille Service de Pneumologie et Oncologie Thoracique, Lille
  - Institut Paoli Calmettes, Marseille
  - Hopital Bichat Claude Bernard, Paris
  - Hopital Tenon, Paris
  - Hopital de Pontchaillou, Rennes
  - CHU Strasbourg - Nouvel Hopital Civil, Strasbourg
  - CHU de Toulouse - Hôpital Larrey, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus, Medizinische Klinik I, Pneumologie MK1-A13, Dresden
  - Asklepios-Fachkliniken Muenchen-Gauting, Gauting
  - Pius-Hospital, Oldenburg
  - Leopoldina-Krankenhaus Medizinische Klinik II, Schweinfurt
  - Klinik Schillerhöhe, Stuttgart
- St. James Hospital, Dublin, Ireland
- Italy (8):
  - Ospedale Clinicizzato SS Annunziata, Chieti, Abruzzo
  - Istituto Nazionale per lo Studio e la Cura dei Tumori Fondazione G. Pascale, Napoli, Campania
  - Ospedale Provinciale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Istituto Nazionale Tumori Regina Elena, Rome, Lazio
  - AZ. Ospedaliera San Giovanni - Addolorata, Rome, Lazio
  - Azienda Ospedaliera Universitaria Pisana - Ospedale Cisanello, Pisa, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
  - A.O.U. INTEGRATA DI VERONA-Ospedale Civile Maggiore Borgo Trento, Verona, Veneto
- Japan (7):
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Osaka International Cancer Institute, Osaka
  - Kansai Medical University Hospital, Osaka
  - Juntendo University Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - National Hospital Organization Yamaguchi - Ube Medical Center, Yamaguchi
- Health Pharma Professional Research, Mexico City, Mexico CITY (federal District), Mexico
- Netherlands (2):
  - NKI/AvL, Amsterdam
  - Maastricht University Medical Center, Maastricht
- Hemato Oncología de Panamá Especializada, Panama City, Panama
- Narod.Inst.Onkol. im. M.Sklodowskiej - Curie-Panst.Inst.Bad, Warsaw, Poland
- IPO do Porto, Porto, Portugal
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (9):
  - Insititut Catala D'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruña, A Coruña, LA Coruna
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital de Madrid Norte Sanchinarro- Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hosp Clinico Univ Lozano Blesa, Zaragoza
- Karolinska Universitetssjukhuset, Solna, Stockholm, Sweden
- UniversitätsSpital Zürich, Zurich, Switzerland
- Turkey (Türkiye) (3):
  - Adana City Hospital, Medical Oncology, Adana
  - Ankara Bilkent City Hospital, Ankara
  - ?zmir Medical Point, Kar?iyaka
- United Kingdom (7):
  - Velindre Cancer Centre, Cardiff
  - Leicester Royal Infirmary, Leicester
  - University College Hospital, London
  - Guys & St Thomas Hospital, London
  - Royal Marsden Hospital, London
  - Christie Hospital Nhs Trust, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing